CLINICAL TRIAL: NCT05089851
Title: A Randomized, Multicenter, Double-blinded, Placebo Controlled, Split-Face Study Evaluating Procedure Pairing of a Peptide Anti-Aging Serum With Onabotulinumtoxin A in the Treatment of Periorbital Facial Wrinkles
Brief Title: Investigation of the Efficacy and Tolerability of a Cosmetic Product With Onabotulinumtoxin A in the Treatment of Facial Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RS-2020-01
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Wrinkles; Photoaging; Fine Lines
Keywords: anti-aging; serum; onabotulinum toxin A; Botox
MeSH Terms: interventions — Botulinum Toxins, Type A; Botulinum Toxins; Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Randomized, Multi-Center, Double-Blinded, Placebo-Controlled, Split-Face
Who Masked: Participant, Investigator
Masking Description: Subjects left and right face (split face) will be randomly assigned to one of the following treatment arms: peptide antiaging serum vs placebo serum. The active and placebo will be placed in the same container and labelled Right and Left. Double blinded study, where the investigator, study subject, and other study personnel involved in the evaluation of the efficacy or safety are blinded to treatment during the twelve week randomization study. The investigational product will be identical in appearance to placebo and both will be packaged in the same container, which will be labelled Right and Left corresponding to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Peptide Antiaging Serum (Active Comparator): Dosage Form: Serum composed of water, thickener, and bioactive ingredients including peptides and antioxidants.
  Frequency of Dosage: Twice daily. Subjects will be asked to pump 1x and apply to assigned facial side (left or right) corresponding to randomization.
  Study Duration: 12 weeks
  Interventions: Procedure: Onabotulinumtoxin A; Combination Product: Facial Cleanser; Combination Product: Facial Moisturizer; Combination Product: Sunscreen
- Placebo Serum (Placebo Comparator): Dosage Form: Serum composed of water and thickener
  Frequency of Dosage: Twice daily. Subjects will be asked to pump 1x and apply to assigned facial side (left or right) corresponding to randomization.
  Study Duration: 12 weeks
  Interventions: Procedure: Onabotulinumtoxin A; Combination Product: Facial Cleanser; Combination Product: Facial Moisturizer; Combination Product: Sunscreen

INTERVENTIONS:
Procedure: Onabotulinumtoxin A — Subjects will receive 20 - 24 units to the crows feet (10 - 12 units per side)
  Other Names: Botulinum Toxin, Allergan
Combination Product: Facial Cleanser — Facial Cleanser to be used by participants twice daily
Combination Product: Facial Moisturizer — Bland moisturizer to be used by study participants after serum twice daily.
Combination Product: Sunscreen — Bland Sunscreen to be used by study participants after serum and moisturizer in the morning. Sunscreen to be reapplied if continuous sun exposure occurs.
  Other Names: Aveeno Face Milk SPF 40+

SUMMARY:
This randomized, multi-center, double-blinded, placebo-controlled, split-face clinical trial was conducted to evaluate the procedure-pairing of OnabotulinumtoxinA with a peptide anti-aging serum to improve facial lines and wrinkles, as well as overall skin texture and radiance of the face after 12 weeks of twice-daily use in female subjects ages 35 - 60 as compared to placebo. A total of 29 subjects completed study participation.

DETAILED DESCRIPTION:
This randomized, multi-center, double-blinded, placebo-controlled, split-face clinical trial was conducted to evaluate procedure pairing of a peptide anti-aging serum with Onabotulinumtoxin A in the treatment of periorbital facial wrinkles when used over the course of 12 weeks by women with moderate to severe crow's feet wrinkles and fine lines, and mild to moderate photoaging.

Efficacy and tolerability will be assessed through clinical grading at baseline, weeks 4, 8 and 12. Efficacy evaluation for wrinkles, fine lines, and skin appearance will be graded at rest and at maximum smile for each side. Investigator and subject tolerability, self-assessment questionnaire and VISIA photography will be completed at baseline, weeks 4, 8 and 12.

A total of 29 subjects completed study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects must be between 35-60 years of age.
2. Female subjects of childbearing potential must be willing to use a form of birth control during the study.
3. Subjects with Fitzpatrick I-VI photo skin type.
4. Subjects must have moderate to severe crow's feet facial wrinkles (score 4-7 on 0-9 scale) using modified Griffith's 10-point scale.
5. Subjects must have moderate to severe crow's feet fine lines (score 4-7 on 0-9 scale) using modified Griffith's 10-point scale.
6. Subjects may have mild to moderate photo-aging (score 3-6 on 0-9 scale) secondary to physiologic aging, hormonal influences, and environmental stressors.
7. Subjects must have no skin disease in the facial area being evaluated.
8. Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation.
9. Subjects must be willing to provide verbal understanding and written informed consent

Exclusion Criteria:

1. Female subjects who are pregnant, breast feeding, or planning a pregnancy.
2. Subjects with severe overall photo damage (score 7-9 on 0-9 scale) as determined by the Investigator.
3. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products or to the botulinum toxin.
4. Subjects who are unwilling or unable to comply with the requirements of the protocol.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-23 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy Grading by Griffith's Scale | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10 point scale. A change in scores at Day 28, Day 56, and Day 84 (+/- 3 days) in comparison to baseline indicates an improvement for the indicated parameter.
  The efficacy parameters will be assessed at rest and at maximum smile and at specific areas on both the left and right sides of the subjects face using a modified Griffith's 10 point scale according to the following numerical definitions (half point scores may be used as necessary to more accurately describe skin conditions)
  0 = None (best possible condition)
  1 to 3 = Mild 4 to 6 = Moderate 7 to 9 = Severe (worst possible condition). The lower the score equates to the best possible outcome.
Tolerability Scores | 12 weeks
  The primary tolerability endpoint will be Investigator Tolerability Assessment of erythema, edema, and dryness. A change in scores or lack of significant change at Day 28, Day 56, and Day 84 in comparison to baseline indicates tolerability / safety of the test material. Four point scale with a lower score indicating a better outcome.
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
Incidence of Adverse Events | 12 weeks
  The primary safety endpoint will be determined by the incidence and severity of adverse events in healthy subjects, including immediate post-procedure and through-out the length of the study.

SECONDARY OUTCOMES:
Self-Assessment Questionnaire | 12 weeks
  The secondary efficacy endpoint will be the Self-Assessment Questionnaire. A change in response values at Day 28, Day 56, and Day 84 indicates and improvement compared to baseline response values. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement / question being asked.
Secondary Tolerability Scores | 12 weeks
  The secondary tolerability endpoint will be Subject Tolerability Assessment of burning, itching, and stinging. A change in scores or lack of significant change at Day 28, Day 56, Day 84, and Day 168 in comparison to baseline indicates tolerability / safety of the test material. Four point scale with a lower score indicating a better outcome.
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Shino Bay Cosmetic Dermatology and Laser Institute, Fort Lauderdale, Florida
  - Infinity Skin Care, Coralville, Iowa
  - Juvly Aesthetics, Columbus, Ohio